CLINICAL TRIAL: NCT06335069
Title: 18F-FDG Versus 68Ga-FAPI-46 as PET Tracer in ER-positive Breast Cancer - a Pilot Study.
Brief Title: 18F-FDG Versus 68Ga-FAPI-46 as PET Tracer in ER-positive Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-508066-15
Record Dates: First submitted 2024-03-11; First posted 2024-03-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Diseases
Keywords: 68Ga-FAPI-46; ER+ breast cancer; PET/CT; PET/MRI
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Intervention Model Description: Single-group, single-center pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional 68Ga-FAPI-46 PET/CT and PET/MRI exam (Experimental): All participating patients will undergo an additional 68Ga-FAPI- 46 PET/CT and 68Ga-FAPI-46 PET/MRI scan prior to their breast cancer treatment.
  Interventions: Diagnostic Test: 68Ga-FAPI-46 PET/CT and 68Ga-FAPI-46 PET/MRI

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 PET/CT and 68Ga-FAPI-46 PET/MRI — All participating patients will undergo an additional 68Ga-FAPI- 46 PET/CT and 68Ga-FAPI-46 PET/MRI scan prior to their breast cancer treatment.

SUMMARY:
The extent of breast cancer is an important prognostic factor in patients diagnosed with this disease. Therefore, adequate staging at diagnosis is a requisite for optimal treatment. In all patients diagnosed with locally advanced breast cancer (LABC), distant staging using 18F-FDG PET/CT is recommended. However, the degree of metabolic uptake in the primary breast tumor is significantly lower in the ER+ subtype compared to HER2+ and triple negative breast cancer (TNBC). As a consequence, a suboptimal 18F-FDG uptake in ER+ breast cancer patients can potentially lead to missed distant metastases. Fibroblast-activating protein inhibitor (FAPI) is a recently developed radiotracer that binds to FAP, a stromal antigen overexpressed in more than 90% of epithelial-derived tumors and their metastases. Previous studies all show 68Ga-FAPI PET/CT to have a higher detection rate compared to 18F-FDG PET/CT. However, all previous studies were performed without considering breast cancer subtype. If the metabolic uptake by 68Ga-FAPI-46 is higher in ER+ breast cancer patients, more lesions will be detected, resulting in a more appropriate treatment for these patients. Therefore, in this pilot study, the investigators aim to compare the diagnostic performance of 18F-FDG with 68Ga-FAPI-46 as PET-tracer in ER+ breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with histopathologically proven ER+ breast cancer.
* Diagnosed with locally advanced (primary tumor >5 cm and/or presence of axillary lymph node metastases) or recurrent breast cancer, or metastatic breast cancer for which 18F-FDG PET/CT or 18F-FDG PET/MRI staging is performed.
* Willing and able to undergo the study procedures.
* Has personally provided written informed consent.

Exclusion Criteria:

* Age <18
* Pregnancy
* Patients with secondary malignancies (except non-melanoma skin cancer)
* No 18F-FDG PET/CT or 18F-FDG PET/MRI scan.
* Contra-indications for PET/MRI such as pacemaker, aneurysm clips, metallic device in their body, severe claustrophobia, and severe obesity
* Chronic inflammatory disease such as rheumatoid arthritis.
* Patients with severe hepatic or renal impairment (eGFR ≤45mL/min/1.73m²)
* Inability to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible to participate in this study.
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To determine essential input parameters for an adequate sample size calculation for a diagnostic study that compares the diagnostic accuracy of 18F-FDG and 68Ga-FAPI-46 as PET tracer in patients with ER+ breast cancer. | Patients will be followed from diagnosis until the additional imaging exams are performed, within 20 working days both PET exams will be performed.
  To investigate the proportion of discordant pairs: the number of lesions detected on 18F-FDG PET but not on 68Ga-FAPI-46 PET and the number of lesions detected on 68Ga-FAPI-46 PET but not on 18F-FDG PET.

SECONDARY OUTCOMES:
To explore the feasibility of taking biopsies in test-positive patients. | Patients will be followed from diagnosis until the additional imaging exams are performed, within 20 working days both PET exams will be performed.
  The proportion of 68Ga-FAPI-46-positive 18F-FDG-negative lesions for which performing a biopsy is not feasible.

OTHER OUTCOMES:
To provide preliminary estimates of the proportion of 68Ga-FAPI-46-positive and 18F-FDG-positive lesions confirmed as true positives and false positives verified by a histological biopsy (gold standard) in patients with ER+ breast cancer. | Patients will be followed from diagnosis until the additional imaging exams are performed, within 20 working days both PET exams will be performed.
  The proportion of 68Ga-FAPI-46-positive lesions and the proportion of 18F-FDG-positive lesions confirmed as true positives or false positives (verified by a biopsy, the gold standard)
To investigate the differences in accuracy between 68Ga-FAPI-46 PET/CT versus 68Ga-FAPI-46 PET/MRI. | Patients will be followed from diagnosis until the additional imaging exams are performed, within 20 working days both PET exams will be performed.
  Diagnostic performance will be compared between both exams (i.e. 68Ga-FAPI-46 PET/CT and 68Ga-FAPI-46 PET/MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No